CLINICAL TRIAL: NCT00411385
Title: Phase3 Study to Evaluate the Efficacy and Safety of AlbuminInterferon in Combination With Ribavirin Compared With Peginterferon in Combination With Ribavirin in Interferon Alfa Naive Subjects With CHC Genotype 2/3.
Brief Title: Efficacy of Albumin Interferon Alfa-2b With Ribavirin Compared to Peg-IFN Alfa-2a With Ribavirin in IFN Naive Patients Geno2/3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1008-C1067; ACHIEVE-2/3
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Hepatitis C; CHC; HepC; Genotype 1; Hepatitis; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis | interventions — peginterferon alfa-2a; Ribavirin

ARMS (3):
- 1 (Experimental): 900 mcg alb-IFN every 2 weeks (12 doses) + Ribavirin 800 micrograms per day
  Interventions: Drug: albumin interferon alfa-2b; Drug: Ribavirin
- 2 (Experimental): 1200 mcg alb-IFN every 2 weeks (12 doses) + Ribavirin 800 micrograms per day
  Interventions: Drug: albumin interferon alfa-2b; Drug: Ribavirin
- 3 (Active Comparator): 180 mcg PEG-IFNx2a every 1 week (24 doses)+ Ribavirin 800 micrograms per day
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: albumin interferon alfa-2b — 900 and 1200 micrograms Albumin Interferon Alpha 2a given subcutaneously once every two weeks for 24 weeks
  Arms: 1; 2
Drug: peginterferon alfa-2a — 180 micrograms Pegasys given subcutaneaously once a week for 24 weeks
  Arms: 3
Drug: Ribavirin — 800mg/day for 24 weeks

SUMMARY:
This is a phase 3, randomized, multi-center study to evaluate the efficacy and safety of albumin interferon alfa-2b (alb-IFN)in combination with ribavirin compared with peginterferon alfa-2a (PEGASYS or PEG-IFNa2a) in combination with ribavirin in subjects with chronic hepatitis C, genotype 2/3 who are IFNa treatment naive.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic hepatitis C.
* Liver biopsy performed within 2 years of Day 0 or during screening.
* Infected with hepatitis C virus genotype 2/3.
* Interferon alfa treatment naïve (ie, have never been treated with an interferon product).
* Subjects are eligible to enter the study if they (or their partners) are not pregnant or nursing, are sterile, or of non childbearing potential, or are willing to practice abstinence or use appropriate birth control methods during the study and for 7 months after the last dose of ribavirin.
* Have compensated liver disease.

Key Exclusion Criteria:

* Decompensated liver disease including those subjects with a past history or presence of ascites, bleeding varices or hepatic encephalopathy.
* History of moderate, severe or uncontrolled psychiatric disease, especially depression, including a history of hospitalization or prior suicidal attempt.
* Positive for human immunodeficiency virus (HIV-1) or hepatitis B surface antigen (HBsAG).
* Clinical diagnosis of other causes of chronic liver disease including but not limited to hepatitis B, autoimmune hepatitis, primary biliary cirrhosis, alcoholic liver disease, hemochromatosis, Wilson's Disease, or alpha 1-antitrypsin deficiency.
* A history of immunologically mediated disease (eg, rheumatoid arthritis, inflammatory bowel disease, moderate/severe psoriasis, sarcoidosis, systemic lupus erythematosus).
* Active seizure disorder within the last 2 years.
* Organ transplant other than cornea and hair transplant.
* Clinically significant hemoglobinopathy (eg, thalassemia, sickle cell anemia).
* Cancer within the last 5 years(with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix).
* Drug or alcohol addiction within the last 6 months. Subjects in a supervised methadone treatment program may be enrolled in the study.
* Received any experimental agent within 28 days prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | Week 48

SECONDARY OUTCOMES:
Rapid virologic response | Week 4
Early virologic response | Week 12
Undetectable HCV RNA | Week 24
Normalization of ALT (a liver enzyme) | Week 48
Quality of life evaluation | Week 48
Safety assessments (physical exams, Ae reporting, lab testing/analysis, HADS and Immunogenicity results) | Througout the entire treatment period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (159):
- United States (28):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Florida-Gainesville, Gainesville, Florida
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - Mayo Clinic Transplant Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - GI of Atlanta, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Johns Hopkins Center for Viral Hepatits, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico, Albuquerque, New Mexico
  - New York Hospital - Cornell, New York, New York
  - Faculty Practice Associates, New York, New York
  - NY Presbyterian Medical Center - Columbia Univ. Med Center, New York, New York
  - Bronx VA Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Alamo Medrical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
- Argentina (5):
  - Unidad de Hepatología, Capital Federal, Buenos Aires
  - Fundación Cidea, Capital Federal, Buenos Aires
  - Hospital Italiano, Capital Federal, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Htal Pcial del Centenario, Rosario, Santa Fe Province
- Australia (15):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital Clinical School of Medicine, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gallipoli Research Foundation and Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Bribane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Hospital, Heidelburg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Belgium (5):
  - CHU Brugmann ULB - site Victor Horta, Brussels
  - UCL, Brussels
  - University Hospital Antwerp, Edegem
  - Ghent University Hospital, Ghent
  - CHU Sart Tilman, Liège
- Brazil (5):
  - Hospital Universitário Professor Edgard Santos - Universidade Federal da Bahia, Salvador, Estado de Bahia
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Universidade Federal de São Paulo - UNIFESP, São Paulo, São Paulo
  - Hospital Heliópolis, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
- Canada (10):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - University of Western Ontario Hospital, London, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- France (10):
  - Hopital Beaujon, Clichy
  - Hopital Henri Mondor, Créteil
  - CHU de Lyon, Hôpital de l'Hôtel Dieu, Lyon
  - Hopital Saint-Joseph, Marseille
  - Hopital de La Source, Orléans
  - Hôpital Saint-Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Haut-Leveque, Pessac
  - CHU Purpan Clinique Dieulafoy, Toulouse
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (11):
  - UH Charite Berlin / Virchow Klinikum, Berlin
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Universitätsklinik Düsseldorf, Düsseldorf
  - UH Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Albert-Ludwigs-Universitaet Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Gutenberg-Universitaet Mainz, Mainz
  - Paracelsus Klinik der Stadt Marl, Marl
- India (5):
  - Dayanand Medical College and Hospital, Ludhiana
  - Jaslok Hospital and Research Centre and Breach Candy Hospital,, Mumbai
  - P. D. Hinduja National Hospital and Medical Research Centre, Mumbai
  - G.B.Pant Hospital, New Delhi
  - Maulana Azad Medical College and Associated Lok Nayak Hospital, New Delhi
- Israel (6):
  - Bnei-Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Malaysia (5):
  - Hospital Alor Setar, Alor Star
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - HUKM, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
- Mexico (3):
  - Hosp. Universitario. Monterrey, Monterrey N.L., CP
  - Instituto Nac. de Cs Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico City
  - Clínica Lomas Altas, Mexico City
- Poland (7):
  - Wojewódzki Szpital Specjalistyczny, Bialystok
  - Niepubliczny Zaklad Opieki Zdrowotnej, Czeladź
  - Wojewódzki Szpital Zespolony, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersytet Medyczny, Lodz
  - Wojewódzki Szpital Zakaźny, Warsaw
  - Przychodnia przy Łowieckie, Wroclaw
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - CGH, Singapore
- South Korea (12):
  - Bundang CHA Hospital, Bundang
  - Kyungpook National University Hospital, Daegu
  - Pusan National University Hospital, Pusan
  - Seoul National University Hospital(Bundang), Seonnam City
  - Severance Hospital(SVR), Seoul
  - Kyunghee University - Medical center, Seoul
  - Samsung Medical Center, Seoul
  - Yongdong Severance Hospital, Seoul
  - Korea University Medical Center(Anam), Seoul
  - Asan Medical Center, Seoul
  - Korea University Medical Center(Guro), Seoul
  - Aju University Hospital, Suwon
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Badalona - Barcelona
  - Hopital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Carlos III, Madrid
  - Complejo Hospitalario Nuestra Señora de Valme, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Universitetssjukhuset MAS, Malmo
  - Karolinska Universitetssjukhuset, Stockholm
- Taiwan (12):
  - TCGH-HL, Hualien City, R.o.c.
  - KMUH, Kaohsiung City, R.o.c.
  - KCGMH, Kaohsiung City, R.o.c.
  - VGH-TC, Taichung, R.o.c.
  - NTUH, Taipei, R.o.c.
  - TSGH, Taipei, R.o.c.
  - CGMH-LK, Taoyuan District, R.o.c.
  - CCH, Changhua
  - CMUH, Taichung
  - NCKUH, Tainan
  - CMMC, Tainan
  - TCGH-TP, Taipei
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai
- Barts and the London NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Bain VG, Yoshida EM, Kaita KD, Swain MG, Heathcote EJ, Garcia A, Moore PA, Yu R, McHutchison JG, Subramanian GM. Dynamics of interferon-specific gene expression in peripheral blood of interferon alfa-naive patients with genotype 1 chronic hepatitis C infection treated with albumin-interferon alfa. Hepatol Res. 2006 Aug;35(4):256-62. doi: 10.1016/j.hepres.2006.04.005. Epub 2006 May 30. PMID 16731032
- [Background] Bain VG, Kaita KD, Yoshida EM, Swain MG, Heathcote EJ, Neumann AU, Fiscella M, Yu R, Osborn BL, Cronin PW, Freimuth WW, McHutchison JG, Subramanian GM. A phase 2 study to evaluate the antiviral activity, safety, and pharmacokinetics of recombinant human albumin-interferon alfa fusion protein in genotype 1 chronic hepatitis C patients. J Hepatol. 2006 Apr;44(4):671-8. doi: 10.1016/j.jhep.2005.12.011. Epub 2006 Jan 30. PMID 16487617
- [Background] S. Zeuzem, , Y. Benhamou, , D. Shouval, , V. Bain, S. Pianko, , R. Flisiak, , M. Grigorescu, , V. Rehak, , E. Yoshida, K. Kaita, , C. Hezode, A.U. Neumann, M. Subramanian, J. McHutchison. Interim (Week 12) Phase 2B Virological Efficacy and Safety Results of albumin interferon alfa-2b Combined with Ribavirin in Genotype 1 Chronic Hepatitis C Infection. EASL, 2006
- [Background] Vinod Rustgi, et al. A Dose-Escalation Study of albumin alfa-Ribavirin in Non-responders to Prior Interferon Based Therapy for Chronic Hepatitis C Infection Phase 2 Dose A Phase 2 Dose-Escalation Study of albumin interferon alfa interferon alfa-2b Combined with 2b Combined with Ribavirin in Non Non-responders to Prior Interferon. EASL, 2006
- [Background] Balan V, Nelson DR, Sulkowski MS, Everson GT, Lambiase LR, Wiesner RH, Dickson RC, Post AB, Redfield RR, Davis GL, Neumann AU, Osborn BL, Freimuth WW, Subramanian GM. A Phase I/II study evaluating escalating doses of recombinant human albumin-interferon-alpha fusion protein in chronic hepatitis C patients who have failed previous interferon-alpha-based therapy. Antivir Ther. 2006;11(1):35-45. PMID 16518958
- [Derived] Nelson DR, Benhamou Y, Chuang WL, Lawitz EJ, Rodriguez-Torres M, Flisiak R, Rasenack JW, Kryczka W, Lee CM, Bain VG, Pianko S, Patel K, Cronin PW, Pulkstenis E, Subramanian GM, McHutchison JG; ACHIEVE-2/3 Study Team. Albinterferon Alfa-2b was not inferior to pegylated interferon-alpha in a randomized trial of patients with chronic hepatitis C virus genotype 2 or 3. Gastroenterology. 2010 Oct;139(4):1267-76. doi: 10.1053/j.gastro.2010.06.062. Epub 2010 Jul 1. PMID 20600017